CLINICAL TRIAL: NCT00125710
Title: Comparative 2-D Tumor Analysis in Familial Gliomas
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: CNS-659
Record Dates: First submitted 2005-07-29; First posted 2005-08-02 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Malignant Glioma
Keywords: cryogenic analysis; oncogenes
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The treatment for patients with malignant brain tumors is disappointing. The disease is incurable and virtually all patients die from their disease. Despite the devastating nature of this illness which affects all age groups, its cause remains unexplained. Family identification with careful clinical and molecular study have led to the discovery of the genes that cause a number of other devastating diseases like retinoblastoma, cystic fibrosis, and Huntington's chorea. The investigators propose to study the genetic changes in patients with familial glioma as a first step in identifying the gene(s) that cause these tumors.

DETAILED DESCRIPTION:
The investigators propose to study the genetic changes in patients with familial glioma as the first step in identifying the gene(s) that cause these tumors. With informed consent, DNAs from tumor and non-tumor tissue, histologic sections, pedigrees and detailed clinical information will be acquired for patients with familial gliomas. A genomic screening methodology named 2D genomic scanning will be used. Differences detected between the tumor and normal tissues (blood, fibroblasts) will identify events occurring in the tumoral process. A comparison of the events in familial and sporadic gliomas will outline some of the pathways suspected to be involved both in tumor initiation and progression. Briefly, DNA fragments are amplified with the polymerase-chain-reaction (PCR) from tumor and normal tissue using primers designed to identify 100 to 1000 random sites within the genome. The PCR primers will hybridize throughout the genome and generate a manageable number of short PCR products that are detected by gel electrophoresis and autoradiography. The PCR for both tumor and constitutional tissues are amplified through 20 to 25 cycles to ensure adequate signal but to avoid entering a non-exponential phase of the PCR amplification. The products are radiolabelled and then run on a standard sequencing gel. The single lane containing labelled PCR products is cut out and then overlaid onto a denaturing grading gel with a 10 to 75% grading of denaturant. The labelled DNA is then separated in the second dimension and the DNA is detected by Southern Transfer to nylon membrane or by gel-drying and direct exposure film. A direct comparison of PCR signals from the tumor and constitutional tissue identifies the loss or gain of signal which reflects the same phenomena within the genome. The isolation and characterization of fragment consistently altered in gliomas will provide the first step in the search for genes responsible in the initiation and progression of gliomas. Because of the collaboration among investigators of different centres in Canada, the current investigators have a unique opportunity to perform the study on the largest collection of familial gliomas in the world. They expect several genomic abnormalities in each tumor. Some of these may be seen in several patients. Data will be analyzed primarily using descriptive statistics, with frequency of genetic abnormalities at different chromosomal locations described.

ELIGIBILITY:
Inclusion Criteria:

* Malignant glioma with a blood relative with history of malignant glioma

Exclusion Criteria:

* Inability to give consent
* Above criteria not met

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 1998-06; Primary Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilson Roa, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada